CLINICAL TRIAL: NCT00006244
Title: Immunotherapy for Autologous/Syngeneic Peripheral Blood Stem Cell (PBSC) Transplant Patients as Treatment for Advanced Multiple Myeloma
Brief Title: Melphalan, Peripheral Stem Cell Transplantation, and Interleukin-2 Followed by Interferon Alfa in Treating Patients With Advanced Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leona Holmberg, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1461.00; NCI-2011-01313 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Interferon-alpha; Interferon Alfa-n3; Introns; Interferon alpha-2; aldesleukin; Interleukin-2; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (immunotherapy) (Experimental): Patients receive melphalan IV over 2-3 hours on day -2 and an infusion of IL-2-treated autologous or syngeneic peripheral blood stem cells on day 0. Beginning on day 0, patients also receive IL-2 IV continuously over 5 days followed by 2 days off. Treatment with IL-2 repeats weekly for 4 weeks. Beginning 1 month later, patients undergo maintenance therapy comprising interferon alfa SC 3 times a week in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: melphalan; Biological: recombinant interferon alfa; Biological: aldesleukin; Procedure: in vitro-treated peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Biological: recombinant interferon alfa — Given SC
  Other Names: Alferon N; alpha interferon; IFN-A; Intron A; Roferon-A
Biological: aldesleukin — Undergo IL2-treated autologous or syngeneic peripheral blood stem infusion
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Procedure: in vitro-treated peripheral blood stem cell transplantation — Undergo IL2-treated autologous or syngeneic peripheral blood stem infusion
  Other Names: in vitro-treated PBPC transplantation; in vitro-treated PBSC; in vitro-treated peripheral blood progenitor cell transplantation; PBPC transplantation, in vitro-treated; peripheral blood progenitor cell transplantation, in vitro-treated

SUMMARY:
This phase II trial studies the effectiveness of melphalan, peripheral stem cell transplantation, and interleukin-2 followed by interferon alfa in treating patients who have advanced multiple myeloma (MM). Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Interleukin-2 (IL2) may stimulate a person's white blood cells to kill multiple myeloma cells. Interferon alfa may interfere with the growth of cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate initial response to therapy, time to disease progression, and overall survival in MM patients treated with melphalan, IL2- incubated peripheral blood stem cells, and sequential IL2.

SECONDARY OBJECTIVES:

I. Evaluate grade 3-4 toxicities encountered by younger (< 56 years old) and older (>56 years old) advanced multiple myeloma patients treated with melphalan, IL2-incubated peripheral blood stem cells, and sequential IL2.

OUTLINE:

Patients receive melphalan intravenously (IV) over 2-3 hours on day -2 and an infusion of IL-2-treated autologous or syngeneic peripheral blood stem cells on day 0. Beginning on day 0, patients also receive IL-2 IV continuously over 5 days followed by 2 days off. Treatment with IL-2 repeats weekly for 4 weeks. Beginning 1 month later, patients undergo maintenance therapy comprising interferon alfa subcutaneously (SC) 3 times a week in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be less than 70 years old
* Patients with advanced Multiple Myeloma that meet the eligibility requirements for mobilization/debulking with Cytoxan/VP-16/G-CSF, Cytoxan/Taxol/G-CSF, or Cytoxan/G-CSF (according to protocol 506.03); if clinically indicated a lower dose of cytoxan than 4g/m2 may be used for mobilization based on the attending's discretion; also, if the patients had previously collected PBSC of sufficient number in the past and meet the other eligibility requirements, they may be entered on this study after approval by the PI
* Patients with advanced Multiple Myeloma that have an identical syngeneic twin for donation of PBSCs
* Patients have advanced Multiple Myeloma if they were diagnosed initially with stage II or III disease or had stage I disease that progressed after initial therapy or failed to respond to therapy
* Syngeneic Donor Inclusion:

  * Donor and patient have adequate documentation that donor and recipient are syngeneic; including ABO typing, HLA typing and VNTR studies
  * Donor > 20 kg
  * Donor meets eligibility to donate according to Standard Practice Guidelines

Exclusion Criteria:

* Patient's age >= 70
* Karnofsky score less than 80
* A left ventricular ejection fraction less than 50%; Patients with congestive heart disease, history of myocardial infarction (MI), coronary artery disease or any arrhythmia history
* Total bilirubin > 1.5 mg/ml (unless history of Gilbert's disease)
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) > 2 x upper limit of normal
* Estimated creatinine clearance < 60 ml/min or creatinine serum > 2.0 mg/dl
* Pregnancy
* Seropositivity for human immunodeficiency virus
* Patients who cannot give informed consent
* Secondary malignancies other than basal cell carcinoma of the skin or carcinoma in situ within the last five years
* History of seizures or requirement for medicines, such as haldol, for controlling mental disorders
* Concurrent need for corticosteroid therapy
* Active connective tissue disease
* Pleural effusion, pericardial effusion or ascites
* Patients allergic to gentamicin
* Patients with positive PCR for hepatitis C or hepatitis B
* Patients with hypersensitivity to E. coli - derived preparations
* Patients with systemic infection at time of IL2 therapy
* Patients who previously have had more than 50% of their pelvic area irradiated
* Patients with pulmonary function tests that show diffusion capacity (corrected) < 60%, and/or forced expiratory volume in 1 second (FEV1) < 65% of predicted

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Immunotherapy Treatment: Patients receive melphalan IV over 2-3 hours on day -2 and an infusion of IL-2-treated autologous or syngeneic peripheral blood stem cells on day 0. Beginning on day 0, patients also receive IL-2 IV continuously over 5 days followed by 2 days off. Treatment with IL-2 repeats weekly for 4 weeks. Beginning 1 month later, patients undergo maintenance therapy comprising interferon alfa SC 3 times a week in the absence of disease progression or unacceptable toxicity.
  melphalan: Given IV
  recombinant interferon alfa: Given SC
  aldesleukin: Undergo IL2-treated autologous or syngeneic peripheral blood stem infusion
  in vitro-treated peripheral blood stem cell transplantation: Undergo IL2-treated autologous or syngeneic peripheral blood stem infusion
Period: Overall Study
Arm/Group | Immunotherapy Treatment
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Immunotherapy Treatment
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: Years] | 53.56 [36.2 to 69.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival in Multiple Myeloma patients treated with melphalan, IL2-incubated peripheral blood stem cells, and sequential IL2 and interferon maintenance.
Time Frame: 12.9 Median Years
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Treatment
Number analyzed (Participants) | 36
Participants | 9

2. Primary Outcome: Initial Response to Therapy
Description: Evaluate initial response to therapy (complete remission, partial remission, stable response, or progression of disease)
Time Frame: Evaluated at Day +84-90 Post-Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Treatment
Number analyzed (Participants) | 36
Participants
  Patients in Complete Remission | 15
  Patients in Partial Remission | 8
  Patients with Stable resposne | 10
  Patients with Disease Progression | 3

3. Primary Outcome: Time to Disease Progression
Time Frame: 12.9 years (median)
Population: Out of 36 patients, 30 have relapsed and they are used to determine this outcome measure.
Measure: Median (Full Range); unit: years
Arm/Group | Immunotherapy Treatment
Number analyzed (Participants) | 30
years | 1.61 [0.12 to 8.96]

4. Primary Outcome: Proportion of Patients Alive and in Remission
Time Frame: 12.9 Median Years
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Treatment
Number analyzed (Participants) | 36
Participants | 4

5. Secondary Outcome: Number of Patients <56 Years Old Experiencing Grade 3-4 Regimen Related Toxicity
Description: Grade 3-4 toxicities by the Bearman common toxicity criteria, encountered by younger (< 56 years old) advanced multiple myeloma patients treated with melphalan, IL2-incubated peripheral blood stem cells, and sequential IL2.
Time Frame: First 100 days post-transplant
Population: Of the 36 patients, 20 patients were <56 years old and these 20 patients are used to determine this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Treatment
Number analyzed (Participants) | 20
Participants | 1

6. Secondary Outcome: Number of Patients ≥56 Years Old Experiencing Grade 3-4 Regimen Related Toxicity
Description: Grade 3-4 toxicities by the Bearman common toxicity criteria, encountered by older (≥56 years old) advanced multiple myeloma patients treated with melphalan, IL2-incubated peripheral blood stem cells, and sequential IL2.
Time Frame: First 100 days post-transplant
Population: Of the 36 patients, 16 patients were ≥56 years old and these 16 are used to determine this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Treatment
Number analyzed (Participants) | 16
Participants | 0

ADVERSE EVENTS:
Arm/Group | Immunotherapy Treatment
All-Cause Mortality (participants affected / at risk) | 27/36
Serious Adverse Events (participants affected / at risk) | 10/36
Other Adverse Events (participants affected / at risk) | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunotherapy Treatment (N=36)
Delayed ANC Engraftment (Blood and lymphatic system disorders) | 1 — Transplant related
Neutropenic fever (Blood and lymphatic system disorders) | 3 — Transplant related
Fever and GI (General disorders) | 1 — Transplant related
Nausea (Gastrointestinal disorders) | 2 — Transplant related One patient also had diarrhea
cardiac event (Cardiac disorders) | 2 — one patient transplant related one patient interferon related
sarcoidosis/failure to thrive (Immune system disorders) | 1 — Interferon related
hypotension (Cardiac disorders) | 1 — Transplant related
mucositis (Gastrointestinal disorders) | 1 — Transplant related
colitis (Gastrointestinal disorders) | 1 — Transplant related
fever (Infections and infestations) | 1 — Transplant related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No